CLINICAL TRIAL: NCT06449287
Title: Strategies to Augment Ketosis: Impact of Exogenous Ketones on Indices of Keto-Adaptation in Obese Subjects on Weight Reducing Diets.
Brief Title: Impact of Exogenous Ketones on Indices of Keto-Adaptation in Obese Subjects on Weight Reducing Diets.
Acronym: STAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017H0395
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Ketogenic Diet; Weight Loss
Keywords: ketones; metabolism; weight loss
MeSH Terms: conditions — Weight Loss; Ketosis | interventions — Diet; Blood Specimen Collection; Ketones; Body Composition; Urinalysis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic Diet (Experimental): Participants will have all their meals prepared in the Instructional Kitchen in the Ohio Union, irrespective of group assignment. They will receive a daily caloric intake equal to 75% of their estimated requirement to maintain weight, which should result in weight loss over the 6-week period. For those in the ketogenic groups, daily macronutrient intake will consist of 35 g of carbohydrates and moderate protein calculated as 1.5 g/kg of reference weight. The remaining caloric intake will consist of fat. A wide range of whole foods will be incorporated into the meals, including non-starchy vegetables, meats, nuts and seeds, oils, cheese, butter, cream, and eggs. The menu will be shared with participants prior to enrolling in the study so they know what to expect in terms of the meal plans.
  Interventions: Other: Diet; Biological: Blood Draw; Biological: Ketone/Glucose Monitoring; Other: Body Composition; Biological: Urine Analysis; Behavioral: Neuropsychological Measures - ANAM
- Ketogenic Diet + Ketone Salt (Experimental): Participants will have all their meals prepared in the Instructional Kitchen in the Ohio Union, irrespective of group assignment. They will receive a daily caloric intake equal to 75% of their estimated requirement to maintain weight, which should result in weight loss over the 6-week period. For those in the ketogenic groups, daily macronutrient intake will consist of 35 g of carbohydrates and moderate protein calculated as 1.5 g/kg of reference weight. The remaining caloric intake will consist of fat. A wide range of whole foods will be incorporated into the meals, including non-starchy vegetables, meats, nuts and seeds, oils, cheese, butter, cream, and eggs. The menu will be shared with participants prior to enrolling in the study so they know what to expect in terms of the meal plans. This group will also be provided a ketone salt supplement to take x2 daily.
  Interventions: Other: Diet; Biological: Blood Draw; Biological: Ketone/Glucose Monitoring; Other: Body Composition; Biological: Urine Analysis; Behavioral: Neuropsychological Measures - ANAM
- Low Fat Diet +Placebo (Active Comparator): The low-fat comparison group will also be provided all their food. Their diet will also be restricted in calories and have the same level of protein, but it will be lower in fat and higher in carbohydrate. The low-fat diet will consist of approximately 25% fat, with the remaining calories coming from carbohydrates (approximately 55% after accounting for protein at around 20%). Added sugars will be kept relatively low (less than 25 g/day) with a focus on unprocessed carbohydrate-rich foods. Saturated fat will be limited to less than 10% of total energy, with a focus on unsaturated fat sources.
  Interventions: Other: Diet; Biological: Blood Draw; Biological: Ketone/Glucose Monitoring; Other: Body Composition; Biological: Urine Analysis; Behavioral: Neuropsychological Measures - ANAM

INTERVENTIONS:
Other: Diet — The diet intervention will start after all baseline testing is complete
Biological: Blood Draw — Blood samples will be collected biweekly.
Biological: Ketone/Glucose Monitoring — Hand-held glucometer will be used daily to monitor dietary intervention adherence.
Other: Body Composition — DEXA Scanning will be done pre-, mid-, and post- intervention.
Biological: Urine Analysis — 24 hour urine collection will be done biweekly.
Behavioral: Neuropsychological Measures - ANAM — The first cognitive assessment will be done via Automated Neuropsychological Assessment Metrics (ANAM). This cognitive battery is a library of computer-based tests of domains including attention, concentration, reaction time, memory, processing speed, decision-making, and executive function.

SUMMARY:
This project will be a three-group controlled 6-wk feeding study where all meals are prepared and provided to obese participants. All participants will be fed a 25% energy-restricted diet. Two diets will be very low in carbohydrate (i.e., ketogenic diets) designed to induce nutritional ketosis and fat loss. Another diet will be low in fat and saturated fat but contain the same total calories. Participants will be randomly assigned to a Ketone Supplement group who are provided an exogenous pre-formed source of beta-hydroxybutyrate (BOHB) or a Control group that only receives the standard ketogenic diet. Randomization will be stratified based on insulin resistance, sex, and body composition to ensure balanced group assignment. Because of timing of recruitment (i.e., after most of the ketogenic groups have already completed the study), the low-fat group will not be randomized. Outcome measurements will be made at various intervals over the 6-wk intervention.

DETAILED DESCRIPTION:
This project will be a three-group controlled 6-wk feeding study where all meals are prepared and provided to obese participants. All participants will be fed a 25% energy-restricted diet. Two diets will be very low in carbohydrate (i.e., ketogenic diets) designed to induce nutritional ketosis and fat loss. Another diet will be low in fat and saturated fat but contain the same total calories. Participants will be randomly assigned to a Ketone Supplement group (n=12) who are provided an exogenous pre-formed source of beta-hydroxybutyrate (BOHB) or a Control group (n=12) that only receives the standard ketogenic diet. Randomization will be stratified based on insulin resistance, sex, and body composition to ensure balanced group assignment. Because of timing of recruitment (i.e., after most of the ketogenic groups have already completed the study), the low-fat group will not be randomized. Outcome measurements will be made at various intervals over the 6-wk intervention. Key outcome variables will include: 1) Markers of Ketosis/Keto-Adaptation: a. Daily measures of BOHB (capillary blood) b. Fasting serum BOHB and total ketones (venous blood) c. Diurnal capillary blood ketones and urinary loss of BOHB and total ketones 2) Energy Balance and Body Composition: a. Body mass (scale) b. Whole body and regional composition (DXA) c. Nitrogen balance (daily nitrogen intake - 24-hr urinary nitrogen loss) d. Resting energy expenditure and substrate oxidation (indirect calorimetry) e. Adiposity (myocardial/epicardial fat, liver fat, visceral fat, skeletal muscle fat by MRI) f. Microbiome (stool collection to observe microbiota and the response to diet alteration) 3) Cognitive and Behavioral: a. Computer-based cognitive function (ANAM) b. Behavioral responses (surveys) 4) Cardio-Metabolic Risk: a. Metabolic panel b. Circulating lipid panel (total cholesterol, LDL-C, HDL-C, TG) c. Glucose, insulin, HOMA

ELIGIBILITY:
Inclusion Criteria:

* BMI >27 and =35 kg/m2

Exclusion Criteria:

* have diabetes, liver, kidney, or other metabolic or endocrine dysfunction, or using diabetic medications.
* Currently consuming a low-carbohydrate diet
* Weight loss of >10% in past 6 months -Currently pregnant or nursing, or planning to become pregnant during the study
* Major psychiatric disorder (e.g., schizophrenia, bipolar disorder)
* Excessive alcohol intake (acute or chronic) defined as average consumption of 3 or more alcohol-containing beverages daily or consumption of more than 14 alcoholic beverages per week

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Daily Ketone/Glucose Monitoring | Up to 6 weeks
  Daily fasting glucose/ketones will be assessed using capillary finger stick lancing. A small drop of blood will be obtained once daily, while fasting, using enzymatic strips fitted for a handheld analyzer (KetoMojo). All the data will be stored in the device's internal memory.
Cholesterol (mg/dl) | up to six weeks
  Fasting venous blood will be collected biweekly to measure cholesterol.
Insulin (mIU/L) | up to six weeks
  Fasting venous blood will be collected biweekly.
Glucose (mg/dL) | up to six weeks
  Fasting venous blood will be collected biweekly.
Lean Mass (kg) | up to six weeks
  DEXA Scanning will be biweekly to assess lean mass
Fat Mass (kg) | up to six weeks
  DEXA Scanning will be biweekly to assess fat mass

SECONDARY OUTCOMES:
Neuropsychological Outcome 1 - Reaction time (Throughput) | up to six weeks
  The first cognitive assessment will be done via Automated Neuropsychological Assessment Metrics (ANAM). Measures SRT by presenting the user with a series of "*" symbols to which they must respond as quickly as possible each time the symbol appears. Results are measured by throughput.
Neuropsychological Outcome 1 - Visual Short Term Memory (Throughput) | up to six weeks
  The first cognitive assessment will be done via Automated Neuropsychological Assessment Metrics (ANAM). Measures verbal short-term memory by having the users memorize a set of characters and then indicate as single characters are presented on the screen whether the character was part of the memory set. Results are measured by throughput.
Neuropsychological Outcome 1 - Spatial Processing (Throughput) | up to six weeks
  The first cognitive assessment will be done via Automated Neuropsychological Assessment Metrics (ANAM). Measures visual spatial skills and mental rotation by having the users compare the equivalence of two 4-bar histograms, the first of which is displayed upright and the second of which is displayed after a 90° rotation either clockwise or counterclockwise. Results are measured by Throughput.
Urine Chemistries | up to 6 weeks
  24 hour urine will be collected biweekly and analyzed for urine chemistries

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Volek, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kackley ML, Brownlow ML, Buga A, Crabtree CD, Sapper TN, O'Connor A, Volek JS. The effects of a 6-week controlled, hypocaloric ketogenic diet, with and without exogenous ketone salts, on cognitive performance and mood states in overweight and obese adults. Front Neurosci. 2022 Sep 30;16:971144. doi: 10.3389/fnins.2022.971144. eCollection 2022. PMID 36248655
- [Result] Belany P, Kackley ML, Zhao S, Kluwe B, Buga A, Crabtree CD, Nedungadi D, Kline D, Brock G, Simonetti OP, Volek JS, Joseph JJ. Effects of Hypocaloric Low-Fat, Ketogenic, and Ketogenic and Ketone Supplement Diets on Aldosterone and Renin. J Clin Endocrinol Metab. 2023 Jun 16;108(7):1727-1739. doi: 10.1210/clinem/dgad009. PMID 36629058
- [Result] Buga A, Kackley ML, Crabtree CD, Bedell TN, Robinson BT, Stoner JT, Decker DD, Hyde PN, LaFountain RA, Brownlow ML, O'Connor A, Krishnan D, McElroy CA, Kraemer WJ, Volek JS. Fasting and diurnal blood ketonemia and glycemia responses to a six-week, energy-controlled ketogenic diet, supplemented with racemic R/S-BHB salts. Clin Nutr ESPEN. 2023 Apr;54:277-287. doi: 10.1016/j.clnesp.2023.01.030. Epub 2023 Feb 4. PMID 36963874